CLINICAL TRIAL: NCT03021993
Title: Phase II Trial of Nivolumab, an Anti-PD-1 Monoclonal Antibody, as a Novel Neoadjuvant Pre-Surgical Therapy for Locally Advanced Oral Cavity Cancer
Brief Title: Trial of Nivolumab as a Novel Neoadjuvant Pre-Surgical Therapy for Locally Advanced Oral Cavity Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 102510
Record Dates: First submitted 2016-12-20; First posted 2017-01-16 (Estimated); Results first posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Oral Cavity SCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Experimental): Nivolumab (OPDIVO) will be administered every two weeks for up to four doses prior to surgery at 3mg/kg
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab will be administered on days 1, 15 and 29. If disease has progressed at day 29, the subject will proceed to surgery. If a response or stable disease is present after the third dose, a fourth dose will be given on day 43, then the subject will proceed to surgery.
  Other Names: OPDIVO

SUMMARY:
The purpose of this study is to look at the effectiveness of nivolumab in patients with oral cavity cancer (OCC) who are about to undergo surgery.

DETAILED DESCRIPTION:
OCC patients who are scheduled for surgery will be given Nivolumab prior to surgery to see if there are any changes in surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed histologically proven locoregional OCSCC without evidence of distant metastases and a clinically determined T-stage of 2-4,

   OR

   Recurrent or persistent histologically proven locoregional OCSCC that was initially treated with surgery alone, and a clinically determined recurrent T-stage of 2-4.

   Note - OCSCC includes the subsites of oral tongue, floor of mouth, gingiva, retromolar trigone, and buccal mucosa.

   Note - To allow sufficient tumor tissue for the immunological analyses, patients with T-stage 1 OCSCC will be excluded
2. Greater than or equal to 18 years of age
3. ECOG performance status of 0 or 1
4. Screening labs must meet the following criteria and must be obtained within 14 days prior to registration:

   * WBC > 2,000/µL
   * Absolute Neutrophil Count >1,500/µL
   * Platelets > 100 X 103/µL
   * Hemoglobin > 9.0 g/dL
   * Serum creatinine < 1.5 X ULN or CrCl > 40mL/min (if using the Cockcroft-Gault formula below):

   Female CrCl = (140 - age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL Male CrCl = (140 - age in years) x weight in kg x 1.00 72 x serum creatinine in mg/dL
   * AST/ALT ≤ 3 x ULN
   * Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
5. Reproductive Status:

WOCBP must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug.

Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception with a failure rate of less than 1% per year for a period of 31 weeks after the last dose of investigational product.

WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 consecutive months of amenorrhea in a woman over 45.

Women of childbearing potential must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to registration Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile) and azoospermic men, are not required to use contraception.

Exclusion Criteria:

1. Prior immunotherapy or treatment with another anti PD 1 agent
2. Prior chemotherapy including Cetuximab or radiation therapy
3. Previous severe hypersensitivity reaction to another monoclonal antibody
4. Women who are pregnant, lactating or expecting to conceive
5. Men who are expecting to father children within the research period
6. Known history of HIV or AIDS
7. Positive test for HBV sAg or HCV antibody indicating acute or chronic infection
8. Concomitant malignancies except cutaneous squamous cell carcinoma or basal cell carcinoma
9. Unresectable primary tumor or regional disease; presence of distant metastases.
10. History of pneumonitis or interstitial lung disease
11. Active, known or suspected autoimmune disease. Note: Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
12. Presence of condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone or equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Neskey, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Knochelmann HM, Horton JD, Liu S, Armeson K, Kaczmar JM, Wyatt MM, Richardson MS, Lomeli SH, Xiong Y, Graboyes EM, Lentsch EJ, Hornig JD, Skoner J, Stalcup S, Spampinato MV, Garrett-Mayer E, O'Quinn EC, Timmers CD, Romeo MJ, Wrangle JM, Young MRI, Rubinstein MP, Day TA, Lo RS, Paulos CM, Neskey DM. Neoadjuvant presurgical PD-1 inhibition in oral cavity squamous cell carcinoma. Cell Rep Med. 2021 Oct 19;2(10):100426. doi: 10.1016/j.xcrm.2021.100426. eCollection 2021 Oct 19. PMID 34755137
- [Derived] Liu S, Knochelmann HM, Lomeli SH, Hong A, Richardson M, Yang Z, Lim RJ, Wang Y, Dumitras C, Krysan K, Timmers C, Romeo MJ, Krieg C, O'Quinn EC, Horton JD, Dubinett SM, Paulos CM, Neskey DM, Lo RS. Response and recurrence correlates in individuals treated with neoadjuvant anti-PD-1 therapy for resectable oral cavity squamous cell carcinoma. Cell Rep Med. 2021 Oct 19;2(10):100411. doi: 10.1016/j.xcrm.2021.100411. eCollection 2021 Oct 19. PMID 34755131
- See also: Xiong et al. BMC Cancer (2020) 20:229 — https://doi.org/10.1186/s12885-020-06726-3
- See also: Knochelmann et al., 2021, Cell Reports Medicine 2, 100426 — https://doi.org/10.1016/j.xcrm.2021.100426

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nivolumab
Started | 17
Completed | 8
Not Completed | 9
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 1
Not completed — enrolled but were not treated | 1
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Arm/Group | Nivolumab
Number analyzed (Participants) | 17
Age, Continuous [Mean (Full Range); unit: years] | 62.6 [47 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate Using Pathological Response
Description: Objective response rate: the sum of patients with either a pCR defined as no invasive and no in situ residuals present in the surgical specimen or partial pathologic response defined at least a 30% reduction in the size of the lesion in the surgical specimen. The reduction in size will be determined by comparing the pretreatment clinical measurements (the sum of the greatest axial measurement obtained with calipers at the time of initial evaluation) with the final pathologic measurements.
Time Frame: Time of surgery (day 36 or day 50)
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab
Number analyzed (Participants) | 12
Participants | 4

2. Secondary Outcome: Level of Treg Cells in Peripheral Blood Using Immunostaining
Description: 1. Levels of Treg cells in pre and post treatment peripheral blood will be evaluated using immunostaining for CD4 and flow cytometric analysis of Foxp3. Differences will be calculated (absolute change and percentage change) between pre and post treatment measures.
Time Frame: Day 1 and time of surgery (day 36 or day 50)
Population: Analysis includes 10 participants with complete pre- and post-treatment samples.
Measure: Mean (Standard Deviation); unit: percentage of treg cells
Arm/Group | Nivolumab
Number analyzed (Participants) | 10
percentage of treg cells
  Pre-treatment | 7.7 (8.4)
  Post-treatment | 9.2 (9.1)

3. Secondary Outcome: Level of Activated T-cells in Peripheral Blood
Description: 2. Levels of activated T-cells in peripheral blood will be assessed using flow cytometry for expression of CD69, IFN γ, T-bet and ICOS in CD4+ cells. Differences will be calculated (absolute change and percentage change) between pre and post treatment measures.
Time Frame: Day 1 and time of surgery (day 36 or day 50)
Population: Analysis includes 10 participants with complete pre- and post-treatment samples.
Measure: Mean (Standard Deviation); unit: percentage of CD8 IFN gamma T-cells
Arm/Group | Nivolumab
Number analyzed (Participants) | 10
percentage of CD8 IFN gamma T-cells
  Pre-treatment | 58 (0.49)
  Post-treatment | 62.2 (0.48)

4. Secondary Outcome: Level of Immune Stimulatory Cytokines in Peripheral Blood
Description: 3. Intratumoral immune activity assessed by levels of immune stimulatory cytokines including IL-2, IFN γ, and IL-12 or inhibitory cytokine, IL10 and TGF-beta, in OCSCC tumor lysates will be measured flow cytometrically by cytokine bead array. Differences will be calculated (absolute change and percentage change) between pre and post treatment measures.
Time Frame: Day 1 and time of surgery (day 36 or day 50)
Population: Analysis includes 10 participants with complete pre- and post-treatment samples.
Measure: Mean (Standard Deviation); unit: percentage of cytokines
Arm/Group | Nivolumab
Number analyzed (Participants) | 10
percentage of cytokines
  Pre-treatment | 26.4 (0.19)
  Post-treatment | 36.7 (0.48)

5. Secondary Outcome: Expression of IFN-gamma in CD4+ Cells
Description: Expression of interferon-gamma in CD4+ cells from peripheral blood of patients following PD-1 inhibition therapy will be compared between pre-treatment peripheral blood samples and post-treatment samples from the same patient.
Time Frame: Day 1 and time of surgery (day 36 or day 50)
Population: Analysis includes 10 participants with complete pre- and post-treatment samples.
Measure: Mean (Standard Deviation); unit: percentage of CD4 positive cells
Arm/Group | Nivolumab
Number analyzed (Participants) | 10
percentage of CD4 positive cells
  Pre-treatment | 20 (12.6)
  Post-treatment | 23.9 (13.5)

6. Secondary Outcome: Expression of Granzyme-B in CD8+ Cells From Peripheral Blood
Description: Expression of Granzyme-B in CD8+ cells from peripheral blood of patients following PD-1 inhibition therapy will be compared between pre-treatment peripheral blood samples and post-treatment samples from the same patient.
Time Frame: Day 1 and time of surgery (day 36 or day 50)
Population: Analysis includes 10 participants with complete pre- and post-treatment samples.
Measure: Mean (Standard Deviation); unit: percentage of CD8 positive cells
Arm/Group | Nivolumab
Number analyzed (Participants) | 10
percentage of CD8 positive cells
  Pre-treatment | 46.7 (15.8)
  Post-treatment | 55.5 (15.7)

7. Secondary Outcome: Expression of CD8+ Cells Expressing Granzyme B (Cytolytic Response) From Peripheral Blood
Description: 2. Expression of CD8+ cells expressing granzyme B (cytolytic response) from peripheral blood of patients following PD-1 inhibition therapy will be compared between pre-treatment peripheral blood samples and post-treatment samples from the same patient.
Time Frame: Day 1 and time of surgery (day 36 or day 50)
Population: Analysis includes 10 participants with complete pre- and post-treatment samples.
Measure: Mean (Standard Deviation); unit: percentage of CD8+cells expressing granz
Arm/Group | Nivolumab
Number analyzed (Participants) | 10
percentage of CD8+cells expressing granz
  Pre-treatment | 34.7 (0.48)
  Post-treatment | 42.6 (0.49)

ADVERSE EVENTS:
Time Frame: 12 months post surgery
Arm/Group | Nivolumab
All-Cause Mortality (participants affected / at risk) | 3/17
Serious Adverse Events (participants affected / at risk) | 1/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab (N=17)
Hypercalcemia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab (N=17)
Painful Swelling In R Submandibular Node (General disorders) | 1 (1)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 1 (1)
Hearing Impaired (Ear and labyrinth disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (8)
Nausea (Gastrointestinal disorders) | 3 (3)
Oral Pain (General disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
muscositis oral (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Thrush (Gastrointestinal disorders) | 1 (1)
Worsened Tongue Pain (Gastrointestinal disorders) | 1 (1)
Xerostomia (Gastrointestinal disorders) | 1 (1)
Numbness Of Tongue (Gastrointestinal disorders) | 1 (1)
Opiod Induced Constipation (Gastrointestinal disorders) | 1 (1)
Tongue Pain (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 4 (4)
Pain (General disorders) | 4 (4)
Edema Face (General disorders) | 2 (2)
Worsened Appetite (General disorders) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1)
Leg Wound Infection At Site Of Graft (Infections and infestations) | 1 (1)
Weight Loss (Investigations) | 5 (5)
Alanine aminotransferase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Right Hand Swollen (Musculoskeletal and connective tissue disorders) | 1 (1)
Stiffness in Arms/Legs (Musculoskeletal and connective tissue disorders) | 1 (1)
T8 Compression Deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Back Spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis Feeling In Thighs And Arms (Musculoskeletal and connective tissue disorders) | 1 (1)
Stiff Neck (Musculoskeletal and connective tissue disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash acneiform (Skin) | 1 (1)
Pruritic Rash Shoulder (Skin) | 1 (1)
Psoriasis (Skin) | 1 (1)
Actinic Keratosis (Skin) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-06): https://cdn.clinicaltrials.gov/large-docs/93/NCT03021993/Prot_SAP_000.pdf
  • Informed Consent Form (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT03021993/ICF_001.pdf